CLINICAL TRIAL: NCT00660426
Title: Phase I Study Of Oxaliplatin, Gemcitabine And Capecitabine In Advanced Gastrointestinal Malignancies And Other Solid Tumors
Brief Title: Study Of Advanced Gastrointestinal Malignancies And Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-1213
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Advanced Gastrointestinal Malignancies; Solid Tumors
Keywords: cancer; gastrointestinal; tumor
MeSH Terms: conditions — Neoplasms | interventions — Oxaliplatin; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level 1 (starting level) (Experimental): Oxaliplatin 85 mg/m2 IV on days 1 and 15.
  Gemcitabine 800 mg/m2 IV on days 1 and 15.
  Capecitabine 600 mg/m2 BID orally on days 1-7 and days 15-21 rounded off to the nearest 150 mg or 500 mg tablet.
  Each cycle is 28 days.
  Interventions: Drug: Oxaliplatin; Drug: Gemcitabine; Drug: Capecitabine
- Dose Level 2 (Experimental): Oxaliplatin 100 mg/m2 IV on days 1 and 15.
  Gemcitabine 800 mg/m2 IV on days 1 and 15.
  Capecitabine 600 mg/m2 BID orally on days 1-7 and days 15-21 rounded off to the nearest 150 mg or 500 mg tablet.
  Each cycle is 28 days.
  Interventions: Drug: Oxaliplatin; Drug: Gemcitabine; Drug: Capecitabine
- Dose Level 3 (Experimental): Oxaliplatin 100 mg/m2 IV on days 1 and 15.
  Gemcitabine 800 mg/m2 IV on days 1 and 15.
  Capecitabine 800 mg/m2 BID orally on days 1-7 and days 15-21 rounded off to the nearest 150 mg or 500 mg tablet.
  Each cycle is 28 days.
  Interventions: Drug: Oxaliplatin; Drug: Gemcitabine; Drug: Capecitabine
- Dose Level 4 (Experimental): Oxaliplatin 100 mg/m2 IV on days 1 and 15.
  Gemcitabine 1000 mg/m2 IV on days 1 and 15.
  Capecitabine 800 mg/m2 BID orally on days 1-7 and days 15-21 rounded off to the nearest 150 mg or 500 mg tablet.
  Each cycle is 28 days.
  Interventions: Drug: Oxaliplatin; Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
Dose escalation of oxaliplatin, gemcitabine and capecitabine in the treatment of patients with advanced gastrointestinal malignancies and other solid tumors.

DETAILED DESCRIPTION:
To define the maximum tolerated dose of oxaliplatin, gemcitabine and capecitabine in the treatment of patients with advanced gastrointestinal malignancies and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histological Diagnosis: Patients must have a histological or cytological proven advanced gastrointestinal or other solid malignancy.
2. Measurable or Evaluable Disease: See RECIST Criteria: www.cancer.gov/dip/RECIST
3. Age: Patients must be 18 years old or older. Because no dosing or toxicity data are currently available on the use of oxaliplatin in patients <18 years of age, children are excluded from this study, but will be eligible for other pediatric Phase I single-agent trials, when available.
4. Performance Status: NCI CTC 0-2.
5. Life Expectancy: >=8 weeks.
6. Recovery from Prior Therapy: Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study and must be without significant systemic illness (e.g. infection). No chemotherapy or radiotherapy may be given within 3 weeks prior to the start of protocol treatment. Patients must have received <= 2 prior chemotherapy regimes.
7. Recovery from Intercurrent Illness: Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
8. Hematological Status: Patients must have adequate bone marrow function which is defined as an absolute neutrophil count >= 1,500/mm³, platelet count >= 100,000/mm³ and hemoglobin >= 9 g/dl.
9. Hepatic Function: Total bilirubin must be <= institutional limit of normal (ULN). Transaminases (SGOT and/or SGPT) must be <= 4 x ULN.
10. Neurological Status: Patients must not have active CNS metastases. Patients with Grade 2 or higher peripheral neuropathy are ineligible due to the potential neurological complications of oxaliplatin therapy.
11. Renal Function: Patients must have adequate renal function defined as serum creatinine <= 2.0 mg/dl or creatinine clearance >= 60 ml/min/1.73m² for patients with creatinine levels above 2.0 mg/dl.
12. Sexually Active Patients: For all sexually active patients, the use of adequate barrier contraception (hormonal or barrier method of birth control) will be required during therapy, prior to study entry and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential. Pregnant and nursing women patients are not eligible.
13. HIV-Positive Patients: Patients receiving anti-retroviral therapy (HAART) for HIV infection are excluded from the study because of possible pharmacokinetic interactions. Appropriate protocols will be offered to patients receiving HAART therapy, when indicated.
14. No known hypersensitivity to oxaliplatin, gemcitabine or capecitabine
15. No pre-existing clinically significant cardiac, hepatic or renal disease.
16. Informed Consent: After being informed of the treatment involved, patients must give written consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.
17. Inclusion of Women and Minorities: Entry to this study is open to both men and women and to all racial and ethnic groups.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-03; Primary Completion 2006-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To define the maximum tolerated dose of oxaliplatin, gemcitabine and capecitabine in the treatment of patients with advanced gastrointestinal malignancies and other solid tumors. | At the end of dose escalation (approximately 18 months)

SECONDARY OUTCOMES:
To determine the dose-limiting toxicity of oxaliplatin, gemcitabine and capecitabine in the treatment of patients with advanced gastrointestinal malignancies and other solid tumors. | Approximately 28 days into treatment
  Completion of 1st cycle
To evaluate the incidence and severity of other toxicities of oxaliplatin, gemcitabine and capecitabine in the treatment of patients with advanced gastrointestinal malignancies and other solid tumors. | 30 days after the end of treatment
To perform a structured neurological assessment and questionnaire and report neurological toxicities of oxaliplatin when used with this combination. | 30 days after end of treatment
To perform correlative pharmacogenomic and pharmacokinetic tests for this novel regimen. | Day 1, 7, 15, and 21
  PKs - expanded cohort only

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu